CLINICAL TRIAL: NCT05550324
Title: IPSC Repository of Pediatric Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Mingtao Zhao (Other)
Responsible Party: Sponsor-Investigator, Mingtao Zhao, Research Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00001788
Record Dates: First submitted 2022-08-08; First posted 2022-09-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Disease; Heart Diseases
Keywords: iPSC
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 6-12mL blood sample depending on age of patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Affected Subjects: The subjects must have the diagnosis of cardiovascular disease
  Interventions: Procedure: Blood draw
- Syndromes associated with Cardiovascular Disease: The subject must have a syndrome associated with cardiovascular disease
  Interventions: Procedure: Blood draw
- Family Members: The subject must be related to an individual in cohort 1 or 2
  Interventions: Procedure: Blood draw
- Controls: The subject is considered a control and does not fall into any of the other cohorts
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — One time intravenous blood draw

SUMMARY:
Obtain blood samples for generation and maintenance of induced pluripotent stem cells (iPSCs) and genomic/DNA sequencing for biomedical research that will improve the understanding and treatment of pediatric cardiovascular disease

DETAILED DESCRIPTION:
Human induced pluripotent stem cells (iPSCs) are a type of pluripotent stem cell which can be generated from easily accessible patient cells, such as peripheral blood mononuclear cells and skin fibroblasts. As iPSCs are epigenetically reprogrammed from somatic cells, they retain all genetic information of the affected patients, thus providing an ideal model for studying the contribution of genetic variation to pediatric cardiovascular disease. In addition, human iPSCs can be differentiated into cardiomyocytes, endothelial cells, smooth muscle cells and cardiac fibroblasts, which are major affected cell types in the heart responsible for cardiovascular disease. Therefore, patient-specific iPSCs possess great promise in modeling pediatric cardiovascular disease, discovering novel drugs and prospective cell regeneration therapy.

The DNA from these patients will be analyzed for point mutations, rare sequence variations, single nucleotide polymorphisms in known cardiac development genes or for chromosomal copy number changes by using state of the art genetic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects must have the diagnosis of cardiovascular disease
2. The subject must have a syndrome associated with cardiovascular disease
3. The subject must be related to an individual in cohort 1 or 2
4. The subject is considered a control and does not fall into any of the other cohorts

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any individual with or without pediatric cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
improve the understanding and treatment of pediatric cardiovascular disease | up to 10 Years
  This is a repository of blood samples that will be used into the future for medical research to improve the understanding and treatment of pediatric cardiovascular disease

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Protected health information will only be shared if subjects consent to future research section of informed consent form